CLINICAL TRIAL: NCT03498664
Title: "Cap-assisted" Endoscopic Mucosal Resection vs Standard "Inject and Cut" Endoscopic Mucosal Resection for Large Colonic "Lateral Spreading Tumors" Treatment: a Randomized Multicentric Study.
Brief Title: EMR-C VS EMR-S in Colonic Lateral Spreading Tumors Treatment (LST)
Acronym: LST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Collaborators: Azienda USL 1 Imperiese (Other); Azienda Ospedaliera Niguarda Cà Granda (Other)
Responsible Party: Principal Investigator, Mario Marini, MD, Director of Gastroenterology and Operative Endoscopy Unit, Santa Maria Alle Scotte Hospital, Siena, Italy., Azienda Ospedaliera Universitaria Senese
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90/2014
Record Dates: First submitted 2018-04-07; First posted 2018-04-17 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Endoscopic Mucosal Resection
Keywords: EMR-C; EMR-S; LST

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMR-C group (Experimental): A plastic cap for mucosectomy (MH-597, Olympus Optical Co., Ltd, Tokyo, Japan) with an outer diameter of 17 mm and a length of 15 mm will be preloaded on the tip of the colonoscope. Inside the distal end of the cap there is a gutter which positions the opened polypectomy snare.
  After submucosal injection, the cap will be applied against the lesion which will be aspirated by "controlled suction", avoiding excessive protrusion of tissue in order not to trap the muscular layer.
  The tissue will then be gripped with the snare and resection will be performed. A specific polypectomy snare which can be adapted into the gutter of the cap will be used (SD-221U-25, Olympus Optical Co., Ltd, Tokyo, Japan).
  Interventions: Device: cap for mucosectomy
- EMR-S group (Active Comparator): The resection will be performed using a standard polypectomy snare, which diameter will be chosen according to the size of the lesion, after lifting the lesion from the underlying layers with a submucosal injection of liquid.
  Interventions: Device: standard snare for polypectomy

INTERVENTIONS:
Device: cap for mucosectomy — endoscopic mucosal resection of colonic lesions with a plastic cap for mucosectomy
  Arms: EMR-C group
Device: standard snare for polypectomy — endoscopic mucosal resection of colonic lesions with standard inject and cut mucosectomy
  Arms: EMR-S group

SUMMARY:
"Lateral Spreading Tumors" (LSTs) are dysplastic lesions whose protrusion within the lumens the colon is not more than twice as compared to the surrounding non-dysplastic mucosa.

They can be divided into two groups:

Granular type (LST-G) and Non Granular type (LST-NG) Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) are currently the most used techniques to resect this type of lesions. Compared to other methods of tissue ablation, EMR allows to carry out the histological evaluation of the resected fragments and ESD of the lesion in toto ("en bloc") EMR is currently the most used technique for removal of LST, but for lesions of ≥ 30 mm the resection is performed "piecemeal", i.e. fragmentary. This can compromise an adequate histological evaluation of the lateral and deep margins of the lesion.

Colonic EMR (EMR-S) is usually performed using a polypectomy snare, after lifting the lesion from the underlying layers with a submucosal injection of liquid (EMR standard or "inject-and-cut"). The aspiration of the lesion inside a plastic cap preloaded on the tip of the colonoscope ("cap-assisted EMR" - EMR-C) is almost exclusively used for the treatment of gastric and esophageal lesions. Its use for lesions of the colon and duodenum has been reported in limited experiences The principal aim of this study is to evaluate the efficacy and the safety of the EMR-C for the removal of large colonic LST-G and LST-NG, comparing it with EMR-S.

DETAILED DESCRIPTION:
Colorectal carcinoma (CRC) is the second cause of death for cancer in industrialized countries, with annual incidence and mortality of about one million and 500.000 case respectively.

It's well known that most of CRC follow the path adenoma-carcinoma: early diagnosis and endoscopic removal of colonic polyps has been proved to be useful in preventing cancer.

Most of colorectal polyps are smaller than 1 cm and can be successfully resected with a standard polypectomy. However, between 0.8% and 5% of patients develop sessile polyps or lesions larger than 20 mm, of which removal can be difficult, requiring high endoscopic experience.

Recent prospective studies report that 7%-36% of CRC have a flat or depressed morphology and are more likely to infiltrate the submucosa compared with polypoid ones.

A univariate analysis has proved that the size of the lesion is the only significant risk factor associated with malignant evolution.

Contrary to sessile polyps (SP) that are protruding lesions without a peduncle and whose base has almost the same dimension of the head, "Lateral Spreading Tumors" (LSTs) are dysplastic lesions whose protrusion within the lumen is not more than twice as compared to the surrounding non-dysplastic mucosa. According to Kudo classification they are larger than 1 cm in size, slightly elevated and extending laterally along the intestinal wall.

They can be divided into two groups (according to Paris Classification, 2005, updated for the colon in Kyoto Classification 2008):

* Granular type (LST-G) characterized by nodular aggregates and sub-classified into homogeneous (0-IIa according to Paris Classification) and mixed nodular (0-IIa, 0-Is + IIa, 0-II+ Is) subtypes.
* Non Granular type (LST-NG) characterized by a non nodular surface and sub-classified into elevated (0-IIa) and pseudo-depressed (0-IIa + 0-IIc, 0-IIc +0- IIa) subtypes.

The risk of developing cancer is different between the two types (57.7% in LST-NG vs 32.7% in LST-G). LST-NG are more likely to invade the submucosa compared to LST-G (14% vs 7%). Within the LST-G group, lesions with a mixed nodular morphology have a greater tendency to infiltrate the submucosa compared to the homogeneous ones.

Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) are currently the most used techniques to resect this type of lesions. Compared to other methods of tissue ablation, EMR allows to carry out the histological evaluation of the resected fragments and ESD of the lesion in toto ("en bloc").

EMR allows the resection of superficial neoplasia of gastro-intestinal tract (GI) confined to the mucosa, in the absence of vascular and/or lymphatic invasion.

ESD compared with EMR allows to remove "en bloc" lesions ≥20 mm in size. It should be preferred for lesions with higher risk of invasiveness or when the removal of the deepest layers or of the whole submucosa is desired, despite the size of the lesion. However, ESD is a complex procedure which requires a long training period and it is associated with higher risk of perforation compared with EMR (6.2% vs 1.3%). Furthermore, ESD requires a longer execution time.

Therefore, EMR is currently the most used technique for removal of LST, but for lesions of ≥ 30 mm the resection is performed "piecemeal", i.e. fragmentary. This can compromise an adequate histological evaluation of the lateral and deep margins of the lesion.

Piecemeal resection increases the risk of residual disease that ranges from 12% to 20% compared with 5% described after "en bloc" removal while the percentage of recurrence reported for polypoid lesions ≥ 20 mm is on average 25% (21) and reaches 55% in some studies.

Colonic EMR is usually performed using a polypectomy snare, after lifting the lesion from the underlying layers with a submucosal injection of liquid (EMR standard or "inject-and-cut"). The aspiration of the lesion inside a plastic cap preloaded on the tip of the colonoscope ("cap-assisted EMR" - EMR-C) is almost exclusively used for the treatment of gastric and esophageal lesions. Its use for lesions of the colon and duodenum has been reported in limited experiences.

The advantage of diagnostic "cap-assisted colonoscopy" (CAC) is the higher chance of reaching cecum even by less experienced endoscopists in a shorter time, with less pain for the patients and a better observation of the mucosa behind the folds and at the flexures. There are not enough concordant data about the percentage of missing lesions, especially if small in size (27, 28). The cap makes the position of the instrument more stable during standard "inject-and-cut" technique (EMR-S), and reduces execution time. However, the realization of the EMR-C for colonic lesions isn't reported (29).

The use of EMR-C in colon is controversial because of the risk of entrapping the muscular layer in the polypectomy snare with risk of perforation.

The advantage of using the cap is represented by the possibility to perform mucosectomy of lesions located in difficult positions (between haustra, near or involving the ileo-caecal valve), thanks to the improved visibility on the operative field.

Our group has reported a 4% of residual disease/recurrence rate, much lower than those reported by other authors who performed EMR-S. We had a perforation and bleeding rate of 0% and 7% respectively vs 0.4% and 11% as reported in literature with EMR-S.

More recently, a study of 134 lesions treated with EMR-C reported a recurrence rate of 1.8% on 82 lesions treated, with a mean of 4.2 months follow-up.

The principal aim of this study is to evaluate the efficacy and the safety of the EMR-C for the removal of large colonic granular and non-granular Lateral Spreading Tumors (LST-G, LST-NG), comparing it with EMR-S.

Patients with colorectal LST-G/NG ≥30 mm will be included. Patients who refuse endoscopic follow up will be excluded from the study. The total enrollment period will be 6 months Endoscopic evaluation in patients without invasive carcinoma will be performed at 3, 6 and 12 months, and then annually Follow-up period will last 12 months from the enrollment of the last patient.

Will be defined as:

Residual lesion: the presence of adenomatous tissue endoscopically visible at follow-up colonoscopies within the first year from EMR.

Recurrent lesion: the presence of adenomatous tissue endoscopically visible after 2 (at 3 and 6 months from EMR) previous negative colonoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years Colonic LST-G/NG () ≥ 30 mm in size. Patients able to undergo all follow up procedures as indicated in the protocol and to provide written informed consent, at least 48 hours before the intervention (reasoned consent).

Exclusion Criteria:

* Presence of sessile polyps Non polypoid lesions 0-III according to Paris Classification Lesions with suspicion of malignancy (rigidity, non-lifting lesions, mucosal fragility, ulceration) Patients unable to provide informed consent Patients with coagulopathy and INR >1.5 (not corrected with replacement therapy, such as enoxaparin).

Patients who have undergone previous attempt of lesion resection (residual disease, local recurrence).

Patients with histological diagnosis of submucosal invading neoplasia who will be sent to surgery and excluded from follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with residual lesions within 12 months. | within 12 months
  Patients with non invasive lesions will undergo follow-up colonoscopies at 3, 6, 12 months and thereafter annually after both EMR-C and EMR-S..
  The presence of adenomatous tissue endoscopically visible at follow-up colonoscopies within the first year from EMR will be considered as residual lesion.
Proportion of patients with recurrence at 12 months. | at 12 months
  The presence of adenomatous tissue endoscopically visible after two previous negative colonoscopies will be defined as recurrence. "

SECONDARY OUTCOMES:
Proportion of patients with early complications within 48 hours and late complications after 48 hours from both endoscopic procedures. | at the time of the procedure, within 48 hours, within 12 months
  Complications are defined as:
  intraprocedural early: within 48 hours; late: after 48 hours from the endoscopic procedure;
  Type of complications:
  Bleeding (intraprocedural, loss of blood from rectum; Perforation (documented with the presence of free air in abdomen by RX and/or CT); Post polipectomy syndrome (abdominal pain with or without fever, without any free air in abdomen reported by radiological investigations)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Marini, MD, Principal Investigator — Gastroenterology and Operative Endoscopy Unit, Santa Maria Alle Scotte Hospital, Siena, Italy.; Massimo Conio, MD, Study Chair — ASL 1 imperiese
Locations (1):
- AOUSenese, Siena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Muto T, Bussey HJ, Morson BC. The evolution of cancer of the colon and rectum. Cancer. 1975 Dec;36(6):2251-70. doi: 10.1002/cncr.2820360944. PMID 1203876
- [Result] Rembacken BJ, Fujii T, Cairns A, Dixon MF, Yoshida S, Chalmers DM, Axon AT. Flat and depressed colonic neoplasms: a prospective study of 1000 colonoscopies in the UK. Lancet. 2000 Apr 8;355(9211):1211-4. doi: 10.1016/s0140-6736(00)02086-9. PMID 10770302
- [Result] Jung M. The 'difficult' polyp: pitfalls for endoscopic removal. Dig Dis. 2012;30 Suppl 2:74-80. doi: 10.1159/000341898. Epub 2012 Nov 23. PMID 23207936
- [Result] Xu MD, Wang XY, Li QL, Zhou PH, Zhang YQ, Zhong YS, Chen WF, Ma LL, Qin WZ, Hu JW, Yao LQ. Colorectal lateral spreading tumor subtypes: clinicopathology and outcome of endoscopic submucosal dissection. Int J Colorectal Dis. 2013 Jan;28(1):63-72. doi: 10.1007/s00384-012-1543-2. Epub 2012 Jul 29. PMID 22842665
- [Result] Tsuda S, Veress B, Toth E, Fork FT. Flat and depressed colorectal tumours in a southern Swedish population: a prospective chromoendoscopic and histopathological study. Gut. 2002 Oct;51(4):550-5. doi: 10.1136/gut.51.4.550. PMID 12235079
- [Result] Saitoh Y, Waxman I, West AB, Popnikolov NK, Gatalica Z, Watari J, Obara T, Kohgo Y, Pasricha PJ. Prevalence and distinctive biologic features of flat colorectal adenomas in a North American population. Gastroenterology. 2001 Jun;120(7):1657-65. doi: 10.1053/gast.2001.24886. PMID 11375947
- [Result] Kim WH, Suh JH, Kim TI, Shin SK, Paik YH, Chung HW, Kim DY, Jeong JH, Kang JK, Kim H, Kim NK. Colorectal flat neoplasia. Dig Liver Dis. 2003 Mar;35(3):165-71. doi: 10.1016/s1590-8658(03)00024-0. PMID 12779070
- [Result] The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon: November 30 to December 1, 2002. Gastrointest Endosc. 2003 Dec;58(6 Suppl):S3-43. doi: 10.1016/s0016-5107(03)02159-x. No abstract available. PMID 14652541
- [Result] Kudo S. Endoscopic mucosal resection of flat and depressed types of early colorectal cancer. Endoscopy. 1993 Sep;25(7):455-61. doi: 10.1055/s-2007-1010367. No abstract available. PMID 8261988
- [Result] Kudo S, Kashida H, Tamura T, Kogure E, Imai Y, Yamano H, Hart AR. Colonoscopic diagnosis and management of nonpolypoid early colorectal cancer. World J Surg. 2000 Sep;24(9):1081-90. doi: 10.1007/s002680010154. PMID 11036286
- [Result] Conio M, Blanchi S, Repici A, Ruggeri C, Fisher DA, Filiberti R. Cap-assisted endoscopic mucosal resection for colorectal polyps. Dis Colon Rectum. 2010 Jun;53(6):919-27. doi: 10.1007/DCR.0b013e3181d95a54. PMID 20485006
- [Result] Uraoka T, Saito Y, Matsuda T, Ikehara H, Gotoda T, Saito D, Fujii T. Endoscopic indications for endoscopic mucosal resection of laterally spreading tumours in the colorectum. Gut. 2006 Nov;55(11):1592-7. doi: 10.1136/gut.2005.087452. Epub 2006 May 8. PMID 16682427
- [Result] Othman MO, Wallace MB. Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) in 2011, a Western perspective. Clin Res Hepatol Gastroenterol. 2011 Apr;35(4):288-94. doi: 10.1016/j.clinre.2011.02.006. Epub 2011 Mar 31. PMID 21458402
- [Result] Saito Y, Fukuzawa M, Matsuda T, Fukunaga S, Sakamoto T, Uraoka T, Nakajima T, Ikehara H, Fu KI, Itoi T, Fujii T. Clinical outcome of endoscopic submucosal dissection versus endoscopic mucosal resection of large colorectal tumors as determined by curative resection. Surg Endosc. 2010 Feb;24(2):343-52. doi: 10.1007/s00464-009-0562-8. Epub 2009 Jun 11. PMID 19517168
- [Result] Moss A, Bourke MJ, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Chen RY, Byth K. Endoscopic mucosal resection outcomes and prediction of submucosal cancer from advanced colonic mucosal neoplasia. Gastroenterology. 2011 Jun;140(7):1909-18. doi: 10.1053/j.gastro.2011.02.062. Epub 2011 Mar 8. PMID 21392504
- [Result] Binmoeller KF, Bohnacker S, Seifert H, Thonke F, Valdeyar H, Soehendra N. Endoscopic snare excision of "giant" colorectal polyps. Gastrointest Endosc. 1996 Mar;43(3):183-8. doi: 10.1016/s0016-5107(96)70313-9. PMID 8857131
- [Result] Woodward TA, Heckman MG, Cleveland P, De Melo S, Raimondo M, Wallace M. Predictors of complete endoscopic mucosal resection of flat and depressed gastrointestinal neoplasia of the colon. Am J Gastroenterol. 2012 May;107(5):650-4. doi: 10.1038/ajg.2011.473. PMID 22552236
- [Result] Khashab M, Eid E, Rusche M, Rex DK. Incidence and predictors of "late" recurrences after endoscopic piecemeal resection of large sessile adenomas. Gastrointest Endosc. 2009 Aug;70(2):344-9. doi: 10.1016/j.gie.2008.10.037. Epub 2009 Feb 27. PMID 19249767
- [Result] Zlatanic J, Waye JD, Kim PS, Baiocco PJ, Gleim GW. Large sessile colonic adenomas: use of argon plasma coagulator to supplement piecemeal snare polypectomy. Gastrointest Endosc. 1999 Jun;49(6):731-5. doi: 10.1016/s0016-5107(99)70291-9. PMID 10343218
- [Result] Mahadeva S, Rembacken BJ. Standard "inject and cut" endoscopic mucosal resection technique is practical and effective in the management of superficial colorectal neoplasms. Surg Endosc. 2009 Feb;23(2):417-22. doi: 10.1007/s00464-008-9983-z. Epub 2008 Sep 20. PMID 18806938
- [Result] Conio M, Repici A, Demarquay JF, Blanchi S, Dumas R, Filiberti R. EMR of large sessile colorectal polyps. Gastrointest Endosc. 2004 Aug;60(2):234-41. doi: 10.1016/s0016-5107(04)01567-6. PMID 15278051
- [Result] Conio M, Blanchi S, Filiberti R, Ruggeri C, Fisher DA. Cap-assisted endoscopic mucosal resection of large polyps involving the ileocecal valve. Endoscopy. 2010 Aug;42(8):677-80. doi: 10.1055/s-0030-1255565. Epub 2010 Jun 30. PMID 20593344
- [Result] Conio M, De Ceglie A, Filiberti R, Fisher DA, Siersema PD. Cap-assisted EMR of large, sporadic, nonampullary duodenal polyps. Gastrointest Endosc. 2012 Dec;76(6):1160-9. doi: 10.1016/j.gie.2012.08.009. Epub 2012 Sep 26. PMID 23021169
- [Result] Park SY, Kim HS, Yoon KW, Cho SB, Lee WS, Park CH, Joo YE, Choi SK, Rew JS. Usefulness of cap-assisted colonoscopy during colonoscopic EMR: a randomized, controlled trial. Gastrointest Endosc. 2011 Oct;74(4):869-75. doi: 10.1016/j.gie.2011.06.005. Epub 2011 Aug 6. PMID 21824612
- [Result] Hewett DG, Rex DK. Cap-fitted colonoscopy: a randomized, tandem colonoscopy study of adenoma miss rates. Gastrointest Endosc. 2010 Oct;72(4):775-81. doi: 10.1016/j.gie.2010.04.030. Epub 2010 Jun 25. PMID 20579648
- [Result] Sanchez-Yague A, Kaltenbach T, Yamamoto H, Anglemyer A, Inoue H, Soetikno R. The endoscopic cap that can (with videos). Gastrointest Endosc. 2012 Jul;76(1):169-78.e1-2. doi: 10.1016/j.gie.2012.04.447. No abstract available. PMID 22726477
- [Result] Buchner AM, Guarner-Argente C, Ginsberg GG. Outcomes of EMR of defiant colorectal lesions directed to an endoscopy referral center. Gastrointest Endosc. 2012 Aug;76(2):255-63. doi: 10.1016/j.gie.2012.02.060. Epub 2012 May 31. PMID 22657404
- [Result] Kashani A, Lo SK, Jamil LH. Cap-assisted Endoscopic Mucosal Resection is Highly Effective for Nonpedunculated Colorectal Lesions. J Clin Gastroenterol. 2016 Feb;50(2):163-8. doi: 10.1097/MCG.0000000000000315. PMID 25811116
- [Result] Jass JR, Sobin LH, Watanabe H. The World Health Organization's histologic classification of gastrointestinal tumors. A commentary on the second edition. Cancer. 1990 Nov 15;66(10):2162-7. doi: 10.1002/1097-0142(19901115)66:103.0.co;2-n. PMID 2171747
- [Result] Schlemper RJ, Riddell RH, Kato Y, Borchard F, Cooper HS, Dawsey SM, Dixon MF, Fenoglio-Preiser CM, Flejou JF, Geboes K, Hattori T, Hirota T, Itabashi M, Iwafuchi M, Iwashita A, Kim YI, Kirchner T, Klimpfinger M, Koike M, Lauwers GY, Lewin KJ, Oberhuber G, Offner F, Price AB, Rubio CA, Shimizu M, Shimoda T, Sipponen P, Solcia E, Stolte M, Watanabe H, Yamabe H. The Vienna classification of gastrointestinal epithelial neoplasia. Gut. 2000 Aug;47(2):251-5. doi: 10.1136/gut.47.2.251. PMID 10896917
- [Result] Belderbos TD, Leenders M, Moons LM, Siersema PD. Local recurrence after endoscopic mucosal resection of nonpedunculated colorectal lesions: systematic review and meta-analysis. Endoscopy. 2014 May;46(5):388-402. doi: 10.1055/s-0034-1364970. Epub 2014 Mar 26. PMID 24671869
- [Derived] Conio M, Manta R, Filiberti RA, Baron TH, Pasquale L, Marini M, De Ceglie A. Cap-assisted EMR versus standard inject and cut EMR for treatment of large colonic laterally spreading tumors: a randomized multicenter study (with videos). Gastrointest Endosc. 2022 Nov;96(5):829-839.e1. doi: 10.1016/j.gie.2022.06.002. Epub 2022 Jun 11. PMID 35697127